CLINICAL TRIAL: NCT06166108
Title: Comparative Evaluation of Magnesium Sulphate Versus Dexamethasone as an Adjuvant to Bupivacaine in Ultrasound Guided Transversus Abdominis Plane Block for Abdominal Hysterectomy as Postoperative Analgesia
Brief Title: Magnesium Sulphate Versus Dexamethasone as an Adjuvant to Bupivacaine in TAP Block for Abdominal Hysterectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Hamdy Mohamed Saleh, Resident physician at the anesthesiology and intensive care unit at Assuit University Hospitals, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAP block in Hysterectomy
Record Dates: First submitted 2023-10-29; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: TAP Block
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M "bupivacaine +normal saline +MgSO4" (Active Comparator): will receive 25 ml volume on each side (20 ml of 0.25% bupivacaine plus 5 ml of normal saline containing 250 mg of MgSO4)
  Interventions: Drug: transversus abdominis plane (TAP) block in Abdominal hysterectomy
- Group D "bupivacaine +normal saline +dexamethasone" (Active Comparator): will receive 25ml volume on each side (20 ml of 0.25% bupivacaine plus 5 ml of normal saline containing 8 mg of dexamethasone)
  Interventions: Drug: transversus abdominis plane (TAP) block in Abdominal hysterectomy

INTERVENTIONS:
Drug: transversus abdominis plane (TAP) block in Abdominal hysterectomy — Comparative evaluation of magnesium sulphate versus dexamethasone as an adjuvant to bupivacaine in ultrasound guided transversus abdominis plane block for Abdominal hysterectomy as postoperative analgesia.

SUMMARY:
The aim of this study is to compare the duration of analgesia obtained by addition of dexamethasone and MgSO4 as adjuvants to bupivacaine in TAP block in patients undergoing Total Abdominal Hysterectomy and to evaluate postoperative analgesic requirements, side effects and level of patient satisfaction.

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is accompanied by an extensive inflammatory response resulting in postoperative discomfort and misery. Such patients require appropriate analgesic treatment to reduce morbidity and complications by blunting autonomic, somatic, and endocrine reflexes. As a result, postoperative analgesia following TAH calls for a multimodal approach.

One of the regional techniques routinely used is the transversus abdominis plane (TAP) block. Its widespread use in abdominal surgeries is due to its technical simplicity and trustworthy analgesia. This block implies administering local anesthetic between the internal oblique muscle and transversus abdominis muscle, which is marked by the lumbar Petit triangle. The primary drawback of single-shot regional blocks is their short duration of action when administered with local anesthetic alone. Several adjuvants, including opioids, alpha 2 agonists, N-methylD-aspartate (NMDA) receptor antagonists, and other drugs, have been utilized to extend the duration of blocks. Opioids are by far the most often used adjuvants, but they accompany a host of unpleasant side effects, such as respiratory depression, drowsiness, nausea, and vomiting. In some studies, using alpha 2 agonists such as Dexmedetomidine and Clonidine has been related to drowsiness and bradycardia.

MgSO4 is an N-methyl-D-aspartate (NMDA) receptor antagonist. It acts by non-competitive antagonism blocking the voltage-dependent ion channels.

Dexamethasone is a highly potent, long-acting glucocorticoid. It inhibits potassium conductance by binding to glucocorticoid receptors which decrease the activity of nociceptive C-fibres and may also prolong the analgesia duration through systemic anti'-inflammatory effects and local vasoconstrictive action.

ELIGIBILITY:
Inclusion Criteria:

* Age 35-70 years
* Female patients
* American society of anesthesiologists (ASA) physical state I-II
* Undergoing Total Abdominal Hysterectomy

Exclusion Criteria:

* Patient's refusal
* Cardio-respiratory conditions
* Convulsions
* Local infection at the block's site
* Bleeding diathesis
* Known allergy to any drugs used in this study

Ages: 35 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Comparasion of postoperative NRS score for 24 hours between the two groups | 24 hours postoperative
  NRS Score: used to assess pain intensity. It is one of the most commonly used pain scales in medicine. The NRS consists of a numeric version of the visual analogue scale. It is a horizontal line with an eleven point numeric range. It is labeled from zero to ten, with zero being an example of someone with no pain and ten being the worst pain possible. This scale can be administered verbally. Rescue analgesia will be nalbuphine 0.1 mg/kg IV when the NRS ≥ 4.

SECONDARY OUTCOMES:
Postoperative hemodynamic parameters | 24 hours postoperative
  Hemodynamic parameters including HR(beat/min), MAP(mmHg), and SpO2(%)
Time required for the first rescue analgesia | 24 hours postoperative
  the time at which the patient demand analgesia will be recorded for each patient
Total amount of rescue analgesic consumption during the first 24 hours postoperatively | 24 hours postoperative
Patient satisfaction score | 24 hours postoperative
  Five-points Likert scale: to evaluate the patients' satisfaction regarding the whole procedure at the end of the postoperative 24 hours. It ranged from (1=very satisfied, 2=satisfied, 3=neither satisfied nor dissatisfied, 4=dissatisfied, 5=very dissatisfied)
PONV intensity by postoperatively | 24 hours postoperative
  The number of attacks of nausea for 24 h will be assessed at 0.5, 1, 2, 4, 6, 12 and 24 h and will be recorded as yes/no. •The number of attacks of vomiting for 24 h will be assessed at 0.5, 1, 2, 4, 6, 12 and 24 h postoperatively and will be recorded as yes/no.

CONTACTS AND LOCATIONS:
Overall Officials: Zain Alabdin Zaree Hassan, Professor, Study Chair — Assiut University; Ahmed Talaat Ahmed, Lecture, Study Director — Assiut University

REFERENCES:
- [Background] Balakrishna KP, Kagalkar ND, Suntan A. Efficacy of Magnesium Sulfate as an Adjuvant to Bupivacaine in Transversus Abdominis Plane Block for Abdominal Hysterectomy Surgeries. Cureus. 2023 Apr 5;15(4):e37156. doi: 10.7759/cureus.37156. eCollection 2023 Apr. PMID 37159770
- [Background] Shambhavi T, Das S, Senapati LK, Padhi PP. Comparative evaluation of bupivacaine with magnesium sulphate and dexamethasone as adjuvants in ultrasound-guided transversus abdominis plane block for open unilateral inguinal hernia surgeries: A randomised controlled trial. Indian J Anaesth. 2023 Apr;67(4):370-375. doi: 10.4103/ija.ija_1091_21. Epub 2023 Apr 10. PMID 37303878